CLINICAL TRIAL: NCT05159193
Title: A Multicentre, Open-label, Randomised Trial of Neoadjuvant Pegylated Liposomal Doxorubicin Plus Cyclophosphamide Sequential Docetaxel Plus Trastuzumab and Pertuzumab Versus Docetaxel Plus Carboplatin Combined With Trastuzumab and Pertuzumab in HER-2 Positive Breast Cancer
Brief Title: Neoadjuvant Treatment Pegylated Liposomal Doxorubicin Plus Cyclophosphamide Sequential Docetaxel Plus Trastuzumab and Pertuzumab Versus Docetaxel Plus Carboplatin Combined With Trastuzumab and Pertuzumab in HER-2 Positive Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DMS-BC-K07
Record Dates: First submitted 2021-11-25; First posted 2021-12-16 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — liposomal doxorubicin; Cyclophosphamide; Trastuzumab; Protons; pertuzumab; Docetaxel; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PLD + C + HP followed by THP (Experimental): pegylated liposomal doxorubicin (PLD) 30 mg/m^2, i.v., d1 + cyclophosphamide (C) 600 mg/m^2, i.v., d1 + trastuzumab (H) 8 mg/kg loading dose, 6 mg/kg maintenance doses, i.v., d1 + pertuzumab (P) 840 mg loading dose, 420 mg maintenance doses, i.v., d1 followed by docetaxel (T) 90~100 mg/m^2, i.v., d1 + trastuzumab (H) 6 mg/kg, i.v., d1 + pertuzumab (P) 420 mg, i.v., d1 q3w, for 4 cycles. After neoadjuvant therapy, patients are required to receive a total of 1 year of treatment with trastuzumab (6mg/kg) combined with pertuzumab (420mg), i.v., d1, q3w, regardless of surgery.
  Interventions: Drug: pegylated liposomal doxorubicin (PLD); Drug: cyclophosphamide (C); Drug: trastuzumab (H); Drug: pertuzumab (P); Drug: docetaxel (T)
- TCbHP (Active Comparator): docetaxel (T) 75 mg/m^2, i.v., d1 + carboplatin (Cb) AUC 6, i.v., d1 + trastuzumab (H) 8 mg/kg loading dose, 6 mg/kg maintenance doses, i.v., d1 + pertuzumab (P) 840 mg loading dose, 420 mg maintenance doses, i.v., d1 q3w, for 6 cycles. After neoadjuvant therapy, patients are required to receive a total of 1 year of treatment with trastuzumab (6mg/kg) combined with pertuzumab (420mg), i.v., d1, q3w, regardless of surgery.
  Interventions: Drug: docetaxel (T); Drug: carboplatin (Cb); Drug: trastuzumab (H); Drug: pertuzumab (P)

INTERVENTIONS:
Drug: pegylated liposomal doxorubicin (PLD) — pegylated liposomal doxorubicin (PLD) 30 mg/m^2, i.v., d1, q3w
  Other Names: duomeisu; Doxorubicin Hydrochloride Liposome Injection
  Arms: PLD + C + HP followed by THP
Drug: cyclophosphamide (C) — cyclophosphamide (C) 600 mg/m^2, i.v., d1, q3w
  Other Names: huanlinxianan
  Arms: PLD + C + HP followed by THP
Drug: trastuzumab (H) — trastuzumab (H) 8 mg/kg loading dose, 6 mg/kg maintenance doses, i.v., d1, q3w
  Other Names: qutuozhudankang
  Arms: PLD + C + HP followed by THP
Drug: pertuzumab (P) — pertuzumab (P) 840 mg loading dose, 420 mg maintenance doses, i.v., d1, q3w
  Other Names: patuozhudankang
  Arms: PLD + C + HP followed by THP
Drug: docetaxel (T) — docetaxel (T) 90~100 mg/m^2, i.v., d1, q3w
  Other Names: duoxitasai
  Arms: PLD + C + HP followed by THP
Drug: docetaxel (T) — docetaxel (T) 75 mg/m^2, i.v., d1, q3w
  Other Names: duoxitasai
  Arms: TCbHP
Drug: carboplatin (Cb) — carboplatin (Cb) AUC 6, i.v., d1, q3w
  Other Names: kabo
  Arms: TCbHP
Drug: trastuzumab (H) — trastuzumab (H) 8 mg/kg loading dose, 6 mg/kg maintenance doses, i.v., d1, q3w
  Other Names: qutuozhudankang
  Arms: TCbHP
Drug: pertuzumab (P) — pertuzumab (P) 840 mg loading dose, 420 mg maintenance doses, i.v., d1, q3w
  Other Names: patuozhudankang
  Arms: TCbHP

SUMMARY:
This is a multicenter, open label, non-inferiority, randomized controlled clinical study.

The aim of this study is to evaluate the efficacy and safety of a pegylated liposomal doxorubicin + cyclophosphamide followed by docetaxel plus trastuzumab and pertuzumab (PLD + C + HP followed by THP) regimen compared with a docetaxel + carboplatin plus trastuzumab and pertuzumab (TCbHP) regimen in the neoadjuvant treatment of HER-2-positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged from 18 to 70 years old;
2. Histologically confirmed as invasive breast cancer and without previous treatment.;
3. HER-2 Positive (defined by IHC 3+ or ISH positive);
4. Tumor > 2cm;
5. Biopsy pathology (FNAB or CNB) diagnosed regional lymph node metastasis within 28 days prior to randomization;
6. Participants must have at least one measurable disease according to RECIST 1.1.
7. Participants with multifocal tumors (more than one tumor confined to the same quadrant as the primary tumor) are eligible provided all discrete lesions are sampled and centrally confirmed as HER2 positive.
8. Operable breast cancer with cT2-cT4/cN1-cN3/cM0, according to the AJCC tumor staging manual (8th Edition).
9. The HR(ER and PR) status of the primary tumor and the expression level of Ki-67 are clear.
10. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
11. LVEF ≥ 55%;
12. Brain natriuretic peptide (BNP) (or N-terminal pro brain natriuretic peptide (NT proBNP)) and cardiac troponin assays were within normal values.
13. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP) and serum total bilirubin are all ≤2 ULN. Serum creatinine ≤ 1.5 ULN.
14. Bone marrow function: white blood cell counts ≥ 3.0x10^9/L, absolute neutrophil counts (ANC) ≥ 1.5x10^9/L, platelets ≥ 100x10^9/L, hemoglobin ≥ 90g/L;
15. Participants had good compliance with the planned treatment and follow-up, understood the study procedures of this study, and signed informed consent form.

Exclusion Criteria:

1. Breast cancer with distant metastasis;
2. Participants with multiple lesions (in different quadrants) or bilateral breast cancer;
3. Participants who have received prior anti-cancer therapy for breast cancer except those participants with a history of breast lobular carcinoma in situ (LCIS) that was surgically managed or ductal carcinoma in situ (DCIS) treated exclusively with mastectomy. In case of prior history of LCIS/DCIS, >5 years must have passed from surgery until diagnosis of current breast cancer;
4. In the past and present, participants with severe cardiac disease or discomfort , including but not limited: 1)High-risk uncontrolled arrhythmia, atrial tachycardia (heart rate > 100/min in resting state), significant ventricular arrhythmia (ventricular arrhythmia) or higher atrioventricular block (second-degree type 2 [Mobitz 2] atrioventricular block or third-degree atrioventricular block); 2)Angina pectoris requiring anti-angina medication; 3)Clinically significant valvular heart disease; 4)ECG showing transmural myocardial infarction; 5)Uncontrolled hypertension (eg systolic blood pressure > 180mm Hg or diastolic blood pressure > 100mmHg); 6)Myocardial infarction; 7)Congestive heart failure;
5. Participants have the following serious illnesses or medical conditions, including but not limited: 1)History of serious neurological or psychiatric disorders, including psychosis, dementia, or epilepsy, that prevent understanding and informed consent; 2)Active uncontrolled infection; 3)Active peptic ulcer, unstable diabetes;
6. A history of other malignancies within the previous 5 years, except for adequately treated carcinoma in situ of the cervix or basal cell carcinoma of the skin;
7. Treatment with any investigational drug within 28 days prior to randomization;
8. Participants who are known to be allergic to the active or other components of the study treatment or have contraindications for surgery;
9. Participants who are pregnant, breastfeeding, or refuse to use adequate contraception prior to study entry and for the duration of study participation;
10. Participants who were judged by the investigator to be unsuitable for this study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Estimated)
Dates: Start 2021-12-20 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate | Within 2 to 5 weeks after completion of neoadjuvant therapy
  The percentage of participants without residual invasive cancer (ypT0/Tis ypN0 in the current AJCC staging system) when the complete resected breast specimen and all sampled regional lymph nodes were evaluated with hematoxylin and eosin staining after completion of systemic neoadjuvant therapy.

SECONDARY OUTCOMES:
Objective response rate (ORR) at the end of neoadjuvant chemotherapy | After the last dose to before surgery or within 21 days
  The number of participants who achieved complete response and partial response at the end of neoadjuvant chemotherapy as a percentage of the overall evaluable participants.
5-year disease-free survival (DFS) rate | 5 years
  DFS is defined as the time from randomization to tumor recurrence or death from any cause. 5-year DFS rate is the percentage of participants with DFS from enrollment through 5 years.
Breast conservation rate at surgery | Within 2 to 5 weeks after completion of neoadjuvant therapy
  Percentage of participants receiving breast-conserving surgery after neoadjuvant therapy.
Number of participants with treatment-related adverse events as assessed by NCI-CTCAE V5.0, including overall and Grade 3/4 adverse events. | 5 years
  Number of participants with treatment-related adverse events as assessed by NCI-CTCAE V5.0, including overall and Grade 3/4 adverse events.
Percentage of Participants with dose reductions of chemotherapy due to Grade 3/4 adverse events as assessed by NCI-CTCAE V5.0 | 1 year
  Percentage of Participants with dose reductions of chemotherapy due to Grade 3/4 adverse events as assessed by NCI-CTCAE V5.0
Percentage of Participants with chemotherapy delay due to Grade 3/4 adverse events as assessed by NCI-CTCAE V5.0 | 1 year
  Percentage of Participants with chemotherapy delay due to Grade 3/4 adverse events as assessed by NCI-CTCAE V5.0
Relative dose intensity (RDI) | 1 year
  RDI=actual dose intensity* / standard dose intensity# actual dose intensity* = drug standard dose (mg/m^2) / weeks of administration per cycle (week) standard dose intensity# = actual standard dose (mg/m^2) / actual dosing weeks (week)

OTHER OUTCOMES:
Subgroup analysis of pathological complete response (pCR) rates based on clinically relevant baseline characteristics | Within 2 to 5 weeks after completion of neoadjuvant therapy
  Subgroup analysis of pathological complete response (pCR) rates based on clinically relevant baseline characteristics
Biomarkers | From before neoadjuvant therapy to surgery
  To explore the biomarkers and mechanisms related to neoadjuvant therapy using high-throughput sequencing technology (NGS), and to screen the patients who are suitable for anthracycline-containing neoadjuvant therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Sunyat-sen Memorial Hospital, Guandong, Guangdong, China

IPD SHARING:
Plan to Share IPD: No